CLINICAL TRIAL: NCT02984566
Title: LARK: Liver Ablative Radiotherapy Utilising Kilovoltage Intrafraction Monitoring (KIM)
Brief Title: Liver Ablative Radiotherapy Utilising Kilovoltage Intrafraction Monitoring (KIM)
Acronym: TROG1703 LARK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG1703 LARK
Record Dates: First submitted 2016-11-23; First posted 2016-12-07 (Estimated); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Liver Cancer
Keywords: Primary liver cancer; Secondary liver cancer; Kilovoltage Intrafraction Monitoring; Stereotactic Ablative Body Radiation
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SABR with or without KIM (Experimental): All patients will receive liver SABR. Kilovoltage Intrafraction Monitoring (KIM) tracking will be trialed during mock treatment. If KIM is successful, it will be used throughout treatment. If unsuccessful, cone beam CT will be used instead.
  Interventions: Device: Kilovoltage Intrafraction Monitoring

INTERVENTIONS:
Device: Kilovoltage Intrafraction Monitoring — KIM is a novel intrafraction real-time tumour localization method. It involves a single gantry-mounted kV x-ray imager acquiring 2D projections of implanted fiducial markers. 3D positions are then reconstructed by maximum likelihood estimation of a 3D probability density function.

SUMMARY:
Primary and secondary liver cancer patients will receive liver SABR with or without KIM intervention.

DETAILED DESCRIPTION:
This is a single arm, phase II, two stage study designed to evaluate cancer targeting accuracy, treatment outcomes and treatment efficiency in 46 patients eligible for SABR for either primary or secondary liver malignancy with the incorporation of KIM.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-1
* Life expectancy >6 months
* Number of lesions: ≤ 3
* Lesion size : < 10 cm for a single lesion (and up to 10 cm cumulative diameter for multiple lesions)
* Child-Pugh A or B7 within 6 weeks prior to study entry
* Unsuitable for RFA or resection or transplant
* Distance from GTV to luminal structures (i.e., oesophagus, stomach, duodenum, small or large bowel) ≥ 10mm
* All blood work obtained within 6 weeks prior to study entry with adequate organ function
* May have had previous surgery, RFA or ethanol injection
* Patient must have been discussed at multidisciplinary tumour board with consensus opinion for SBRT

Exclusion Criteria:

* HCC/cholangiocarcinoma with evidence of metastatic disease including nodal or distant metastases
* Metastatic disease with complete liver disease response to first-line chemotherapy (i.e. no target for SBRT)
* Previous radiation to the liver (including SIRTEX)
* Untreated HIV or active hepatitis B/C
* On systemic antineoplastic drug therapy within 7 days before inclusion
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Difference in accumulated patient dose distribution with and without KIM | 15-60 minutes (time of individual fraction delivery)
  Isodose distributions and dose volume histograms for each session will be calculated with KIM corrections as treated, and estimated without KIM corrections. The planning CT scan will be used for this assessment

SECONDARY OUTCOMES:
Difference in treatment time with and without KIM | 15-60 minutes (time of individual fraction delivery)
  The time taken for the KIM treatments compared with the time taken for similar treatments from previous patients, accounting for the difference in the time and number of patient images acquired and the time taken to adjust the patient's position during treatment
Difference in imaging dose with and without KIM | 15-60 minutes (time of individual fraction delivery)
  The KIM procedure adds radiation dose with the kilovoltage images. However, there may be fewer volumetric cone beam computed tomography (CBCT) scans acquired. This difference in dose will be estimated and analysed
Difference in PTV margins with and without KIM | 15-60 minutes (time of individual fraction delivery)
  The clinical target volume (CTV) to planning target volume (PTV) margin with and without KIM will be recorded and analysed.
Difference in accumulated patient dose distribution with and without KIM based on the intra-treatment CBCT scans | 15-60 minutes (time of individual fraction delivery)
  Isodose distributions and dose volume histograms for each session will be calculated with KIM corrections as treated, and estimated without KIM corrections. The intratreatment CBCT scans will be used for this assessment.
Change in dose when using KIM with and without using MLC tracking | 15-60 minutes (time of individual fraction delivery
  Difference between dose delivered using KIM with or without MLC tracking
Proportion of local failures at two years for patients treated | 2 years
  Proportion of local failures at two years for patients treated as assessed using modified RECIST criteria
The proportion of grade 3 or higher toxicities | 2 years
  The proportion of grade 3 or higher toxicities, assessed using CTCAE v4.03
Patient-reported quality of life as measured by the European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Core-30 (EORTC QLQ-C30) | 2 years
  To compare change in Quality of Life, as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQ-C30 (Version 3)) from baseline at completion of radiation therapy and at 6 weeks, 3, 6, 12, 18 and 24 months post-radiation therapy. The EORTC QLQ-C30 (Version 3) uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Half points are not allowed. The range is 3. For the raw score, less points are considered to have a better outcome. The EORTC QLQ-C30 (Version 3) uses for the questions 29 and 30 a 7-points scale. The scale scores from 1 to 7: 1 ("very poor") to 7 ("excellent"). The questionnaire will be self-administered and will be given in patient's mother tongue.
Patient-reported quality of life as measured by the European Organization for Research and Treatment of Cancer Quality-of-Life-Questionnaire-Hepatocellular Carcinoma 18 Module (EORTC QLQ-HCC18) | 18 months
  To compare change in Quality of Life related to hepatocellular carcinoma (HCC) as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Hepatocellular Carcinoma 18 Module (EORTC QLQ-HCC) from baseline at completion of radiation therapy and at 6 weeks, 3, 6, 12 and 18 months post-radiation therapy. The questionnaire will be self-administered and will be given to patients proficient in English. EORTC-QLQ-HCC18: includes HCC-specific symptoms or problems. Questions used 4-point Likert scale from 1 to 4: 1 ("Not at all"), 2 ("A little"), 3 ("Quite a bit") and 4 ("Very much"). Scores averaged and transformed to 0-100 scale. High score for functional scale=high/healthy level of functioning. High score for single item=high level of symptomatology/problems.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wang, Dr, Principal Investigator — Westmead Hospital
Locations (4):
- Australia (4):
  - Nepean Hospital, Penrith, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available to researchers upon request, once evidence of ethical approval has been provided.

REFERENCES:
- [Derived] Lee YYD, Nguyen DT, Moodie T, O'Brien R, McMaster A, Hickey A, Pritchard N, Poulsen P, Tabaksblat EM, Weber B, Worm E, Pryor D, Chu J, Hardcastle N, Booth J, Gebski V, Wang T, Keall P. Study protocol of the LARK (TROG 17.03) clinical trial: a phase II trial investigating the dosimetric impact of Liver Ablative Radiotherapy using Kilovoltage intrafraction monitoring. BMC Cancer. 2021 May 3;21(1):494. doi: 10.1186/s12885-021-08184-x. PMID 33941111